CLINICAL TRIAL: NCT05262387
Title: Effectiveness of a Basal Rate Reduction With LyumjevTM Versus Humalog® on the Protection From Exercise-Induced Hypoglycemia in Individuals With Type 1 Diabetes on Continuous Subcutaneous Insulin Infusion
Brief Title: A Study of LY900014 (Lyumjev) Versus Insulin Lispro (Humalog) in Participants With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17278; I8B-MC-ITSU (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-02-24; First posted 2022-03-02 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Lyumjev; Humalog®; Insulin lispro; Exercise; Continuous Subcutaneous Insulin Infusion; Glycemic control; Hypoglycemia; Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Treatment Sequence 1: ADBC (Experimental): Period 1: Lyumjev with 50% basal rate reduction (Treatment A)
  Period 2: Humalog with 100% basal rate reduction (Treatment D)
  Period 3: Lyumjev with 100% basal rate reduction (Treatment B)
  Period 4: Humalog with 50% basal rate reduction (Treatment C)
  Participants received their assigned treatments in each of the above treatment period on Day 1 subcutaneously.
  Interventions: Drug: Lyumjev with 50% basal rate reduction; Drug: Humalog with 50% basal rate reduction; Drug: Humalog with 100% basal rate reduction; Drug: Lyumjev with 100% basal rate reduction
- Treatment Sequence 2: BACD (Experimental): Period 1: Lyumjev with 100% basal rate reduction (Treatment B)
  Period 2: Lyumjev with 50% basal rate reduction (Treatment A)
  Period 3: Humalog with 50% basal rate reduction (Treatment C)
  Period 4: Humalog with 100% basal rate reduction (Treatment D)
  Participants received their assigned treatments in each of the above treatment period on Day 1 subcutaneously.
  Interventions: Drug: Lyumjev with 50% basal rate reduction; Drug: Humalog with 50% basal rate reduction; Drug: Humalog with 100% basal rate reduction; Drug: Lyumjev with 100% basal rate reduction
- Treatment Sequence 3: CBDA (Experimental): Period 1: Humalog with 50% basal rate reduction (Treatment C)
  Period 2: Lyumjev with 100% basal rate reduction (Treatment B)
  Period 3: Humalog with 100% basal rate reduction (Treatment D)
  Period 4: Lyumjev with 50% basal rate reduction (Treatment A)
  Participants received their assigned treatments in each of the above treatment period on Day 1 subcutaneously.
  Interventions: Drug: Lyumjev with 50% basal rate reduction; Drug: Humalog with 50% basal rate reduction; Drug: Humalog with 100% basal rate reduction; Drug: Lyumjev with 100% basal rate reduction
- Treatment Sequence 4: DCAB (Experimental): Period 1: Humalog with 100% basal rate reduction (Treatment D)
  Period 2: Humalog with 50% basal rate reduction (Treatment C)
  Period 3: Lyumjev with 50% basal rate reduction (Treatment A)
  Period 4: Lyumjev with 100% basal rate reduction (Treatment B)
  Participants received their assigned treatments in each of the above treatment period on Day 1 subcutaneously.
  Interventions: Drug: Lyumjev with 50% basal rate reduction; Drug: Humalog with 50% basal rate reduction; Drug: Humalog with 100% basal rate reduction; Drug: Lyumjev with 100% basal rate reduction

INTERVENTIONS:
Drug: Lyumjev with 50% basal rate reduction — Administered SC.
  Other Names: LY900014
Drug: Humalog with 50% basal rate reduction — Administered SC.
  Other Names: Insulin Lispro
Drug: Humalog with 100% basal rate reduction — Administered SC.
  Other Names: Insulin Lispro
Drug: Lyumjev with 100% basal rate reduction — Administered SC.
  Other Names: LY900014

SUMMARY:
This study will be conducted in participants with type 1 diabetes mellitus on continuous subcutaneous insulin infusion (CSII) or pump therapy to evaluate the effect of LY900014 (Lyumjev) on blood sugar levels during exercise using different approaches on basal rate reduction and following a test meal compared to insulin lispro (Humalog). The study may last up to approximately 10 weeks and may include up to 7 visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants with type 1 diabetes
* Body mass index (BMI) between 18.5 and 29.0 kilograms per square meter (kg/m²), inclusive
* Hemoglobin A1c (HbA1c) less than or equal to 8.5 percent (%)
* Using CSII and stable insulin regimen for at least 6 months prior to inclusion into the trial
* Able to undergo at least 1 hour of moderate-intensity exercise

Exclusion Criteria:

* Are currently participating or recently participated in a clinical trial or any other type of medical research judged to be incompatible with this study
* Have a blood loss of more than 500 milliliters (mL) within the last month
* Have known allergies to insulin lispro, related compounds or any components of the study drug formulation
* Have previously participated or withdrawn from this study
* Have or used to have health problems or medical test results that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Participants who have an abnormal blood pressure and/or pulse rate
* Participants with clinically significant cardiac or pulmonary disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- LMC Clinical Research Inc. (Bayview), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized to 4 treatment sequences (ADBC, BACD, CBDA, and DCAB), with each sequence having 4 periods where participants were crossed over between the periods. A washout period of at least 3 days was maintained between each treatment period.
Period: Treatment Period 1
Arm/Group | Treatment Sequence 1: ADBC | Treatment Sequence 2: BACD | Treatment Sequence 3: CBDA | Treatment Sequence 4: DCAB
Started | 6 | 6 | 7 | 6
Received at Least 1 Dose of Study Drug | 6 | 6 | 7 | 6
Completed | 6 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Treatment Sequence 1: ADBC | Treatment Sequence 2: BACD | Treatment Sequence 3: CBDA | Treatment Sequence 4: DCAB
Started | 6 | 6 | 7 | 6
Completed | 6 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Treatment Sequence 1: ADBC | Treatment Sequence 2: BACD | Treatment Sequence 3: CBDA | Treatment Sequence 4: DCAB
Started | 6 | 6 | 7 | 6
Completed | 6 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | Treatment Sequence 1: ADBC | Treatment Sequence 2: BACD | Treatment Sequence 3: CBDA | Treatment Sequence 4: DCAB
Started | 6 | 6 | 7 | 6
Completed | 6 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- All Participants: Participants received Lyumjev with 50% basal rate reduction (Treatment A) or Lyumjev with 100% basal rate reduction (Treatment B) or Humalog with 50% basal rate reduction (Treatment C) or Humalog with 100% basal rate reduction (Treatment D) subcutaneously on Day 1 in Treatment Period 1 to 4 as per assigned randomized treatment sequence. A washout period of at least 3 days was maintained between all the treatment periods.
Arm/Group | All Participants
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 25

OUTCOME MEASURES:

1. Primary Outcome: Pharmacodynamics (PD): Change in Plasma Glucose (PG) From the Start to the End of Exercise
Description: Changes in PG from the start (0 minute) to end of exercise (60 minutes) were analyzed using a mixed-effect model. The model included treatment (Lyumjev with 50% basal reduction, Lyumjev with 100% basal reduction, Humalog with 50% basal reduction, and Humalog with 100% basal reduction), sequence, period, timepoint, treatment-by-timepoint interaction as fixed effects, and participant-within-sequence as a random effect.
Time Frame: Start (0 minute) to end of exercise (60 minutes)
Population: All participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: milligram per Deciliter (mg/dL)
Groups:
- Lyumjev With 50% Basal Rate Reduction: Participants from all the randomly assigned treatment sequence who received, Lyumjev with 50% basal rate reduction (treatment A), subcutaneously.
- Lyumjev With 100% Basal Rate Reduction: Participants from all the randomly assigned treatment sequence who received, Lyumjev with 100% basal rate reduction (treatment B), subcutaneously.
- Humalog With 50% Basal Rate Reduction: Participants from all the randomly assigned treatment sequence who received, Humalog with 50% basal rate reduction (treatment C), subcutaneously.
- Humalog With 100% Basal Rate Reduction: Participants from all the randomly assigned treatment sequence who received, Humalog with 100% basal rate reduction (treatment D), subcutaneously.
Arm/Group | Lyumjev With 50% Basal Rate Reduction | Lyumjev With 100% Basal Rate Reduction | Humalog With 50% Basal Rate Reduction | Humalog With 100% Basal Rate Reduction
Number analyzed (Participants) | 25 | 25 | 25 | 25
milligram per Deciliter (mg/dL) | -26.8 (37.3) | -46.9 (31.5) | -39.0 (38.8) | -60.5 (39.1)
Statistical Analysis 1: Comparison: Lyumjev With 50% Basal Rate Reduction vs Humalog With 50% Basal Rate Reduction; Test type: Other; p = 0.0494, Mixed Models Analysis; Mean Difference (Final Values) = 9.32, 90% CI 2-sided [1.52 to 17.1]
Statistical Analysis 2: Comparison: Lyumjev With 100% Basal Rate Reduction vs Humalog With 100% Basal Rate Reduction; Test type: Other; p = 0.0028, Mixed Models Analysis; Mean Difference (Final Values) = 14.1, 90% CI 2-sided [6.38 to 21.9]

2. Secondary Outcome: Pharmacodynamics (PD): Change From Baseline in Area Under the Concentration Versus Time Curve From Time 0 to 4 Hours [AUC(0-4)] of Postprandial Plasma Glucose (PPG) Post Mixed-Meal Tolerance Test (MMTT)
Description: The outcome measure was analyzed using a mixed-effect model. The model included treatment (Lyumjev with 50% basal reduction, Lyumjev with 100% basal reduction, Humalog with 50% basal reduction, and Humalog with 100% basal reduction), sequence, and period as fixed effects, and participant-within-sequence will be included as a random effect.
Time Frame: Baseline (0-hour time point prior of the MMTT), 4 hour post-meal MMTT
Population: All participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: milligrams*hour per deciliter (mg*h/dL)
Arm/Group | Lyumjev With 50% Basal Rate Reduction | Lyumjev With 100% Basal Rate Reduction | Humalog With 50% Basal Rate Reduction | Humalog With 100% Basal Rate Reduction
Number analyzed (Participants) | 25 | 25 | 25 | 25
milligrams*hour per deciliter (mg*h/dL) | 247 (121) | 257 (145) | 202 (188) | 262 (129)
Statistical Analysis 1: Comparison: Lyumjev With 50% Basal Rate Reduction vs Humalog With 50% Basal Rate Reduction; Test type: Other; p = 0.1998, Mixed Models Analysis; Mean Difference (Final Values) = -44.5, 90% CI 2-sided [-102 to 12.8]
Statistical Analysis 2: Comparison: Lyumjev With 100% Basal Rate Reduction vs Humalog With 100% Basal Rate Reduction; Test type: Other; p = 0.9041, Mixed Models Analysis; Mean Difference (Final Values) = 4.16, 90% CI 2-sided [-53.1 to 61.4]

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 43
Description: All participants who received at least 1 dose of study drug.
Arm/Group | Lyumjev With 50% Basal Rate Reduction | Lyumjev With 100% Basal Rate Reduction | Humalog With 50% Basal Rate Reduction | Humalog With 100% Basal Rate Reduction
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 4/25 | 2/25 | 3/25 | 4/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lyumjev With 50% Basal Rate Reduction (N=25) | Lyumjev With 100% Basal Rate Reduction (N=25) | Humalog With 50% Basal Rate Reduction (N=25) | Humalog With 100% Basal Rate Reduction (N=25)
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Medical device site pain (General disorders) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT05262387/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/87/NCT05262387/SAP_001.pdf